CLINICAL TRIAL: NCT02601378
Title: A Phase I, Multi-center, Open-label, Study of LXS196, an Oral Protein Kinase C Inhibitor, in Patients With Metastatic Uveal Melanoma
Brief Title: A Phase I Study of LXS196 in Patients With Metastatic Uveal Melanoma.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The combination part of the study was terminated early due to business reasons
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLXS196X2101
Record Dates: First submitted 2015-11-06; First posted 2015-11-10 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Uveal Melanoma
Keywords: Uveal melanoma; Metastatic uveal melanoma; Phase I; LXS196; PKC inhibitor; HDM201; HDM2 inhibitor; dose escalation
MeSH Terms: conditions — Uveal Melanoma | interventions — siremadlin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LXS196 as a single agent (Experimental): About 68 patients will be enrolled in dose escalation and expansion
  Interventions: Drug: LXS196
- LXS196 in combination with HDM201 (Experimental): about 44 patients to be enrolled in dose escalation and expansion
  Interventions: Drug: LXS196 and HDM201

INTERVENTIONS:
Drug: LXS196 — LXS196 as a single agent
  Arms: LXS196 as a single agent
Drug: LXS196 and HDM201 — LXS196 in combination with HDM201
  Arms: LXS196 in combination with HDM201

SUMMARY:
This study was to characterize the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and preliminary anti-tumor activity of LXS196 as a single agent and in combination with HDM201 in patients with metastatic uveal melanoma.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female patients ≥18 years of age
* Diagnosis of uveal melanoma with histological or cytological confirmed metastatic disease. Disease must be treatment naive or have progressed (radiologically or clinically) on most recent therapy.
* Willingness to provide newly obtained tumor tissue at baseline and on treatment unless contraindicated by medical risk in the opinion of the treating physician.
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as >10 mm with CT scan.
* ECOG performance status ≤ 1

Key Exclusion Criteria:

* Malignant disease other than that being treated in this study.
* Symptomatic or untreated CNS metastases or spinal cord compression. Brain metastasis must be stable with verification by imaging .
* Impaired cardiac function or clinically significant cardiac diseases
* History of thromboembolic or cerebrovascular events within the last 6 months, including transient ischemic attack, cerebrovascular accident, deep vein thrombosis, or pulmonary embolism (applicable to combination part only).
* Patients who are receiving treatment with medications that cannot be discontinued prior to study entry and that are considered to be any of the following:
* known and possible risk for QT prolongation
* known to be strong inducers or inhibitors of CYP3A4/5 (for single agent part); known to be moderate to strong inducers or inhibitors of CYP3A4/5 (for combination part)
* known to be inducers or inhibitors of P-gp
* known to be substrates of CYP3A4/5 and P-gp with a narrow therapeutic index
* Patients with abnormal laboratory values, defined as any of the following:
* AST or ALT > 3 times ULN, AST or ALT > 5 times ULN for patients with liver metastases.
* Total bilirubin > 1.5 x ULN, except for patients with Gilbert's syndrome who are excluded if total bilirubin > 3.0 x ULN or direct bilirubin > 1.5 x ULN.
* Absolute neutrophil count (ANC) ≤ 1.5 x109/L.
* Platelets ≤ 100 x 109/L.
* Hemoglobin (Hgb) ≤ 90 g/L (9 g/dL).
* Creatinine > 1.5 x ULN
* Patients receiving live vaccines due to the expected bone marrow toxicity (applicable to combination part only).
* Patients treated with growth factors targeting the myeloid lineage (e.g. G-CSF, GM-CSF and M-CSF) within 2 weeks of starting study treatment. (applicable to combination part only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) (Dose escalation only) | Cycle 1 in dose escalation
  cycle = 28 days
Incidence and severity of adverse events and serious adverse events, including changes in laboratory parameters, vital signs and ECGs graded as per NCI CTCAE version 4.03 (All patients) | Continuously throughout the study until 30 days after treatment discontinuation
Dose interruptions, reductions and dose intensity | Continuously throughout the study until 30 days after treatment discontinuation

SECONDARY OUTCOMES:
Overall response rate (ORR) per RECIST version 1.1 criteria | From baseline, every 2 cycles until cycle 11, then every 3 cycles afterwards until disease progression or withdrawal of consent up to 12 months
Plasma LXS196 concentration-time profiles as a single agent | Cycle 1 Day 1, 2, 3, 15; Cycle 2, 3, 4, 5 and 6 Day1
Modulation of signaling molecules downstream of PKC | Baseline and Cycle 1 Day 15
Progression free survival (PFS) per RECIST version 1.1 criteria | From baseline, every 2 cycles until cycle 11, then every 3 cycles afterwards until disease progression or withdrawal of consent up to 12 months
Plasma PK parameters of LXS196 as a single agent:AUC | Cycle 1 Day 1, 2, 3, 15; Cycle 2, 3, 4, 5 and 6 Day1
Plasma PK parameters of LXS196 as a single agent: Cmax | Cycle 1 Day 1, 2, 3, 15; Cycle 2, 3, 4, 5 and 6 Day1
Plasma PK parameters of LXS196 as a single agent: Tmax | Cycle 1 Day 1, 2, 3, 15; Cycle 2, 3, 4, 5 and 6 Day1
Plasma PK parameters of LXS196 as a single agent: t1/2 | Cycle 1 Day 1, 2, 3, 15; Cycle 2, 3, 4, 5 and 6 Day1
Plasma PK parameters of LXS196 as a single agent: Racc | Cycle 1 Day 1, 2, 3, 15; Cycle 2, 3, 4, 5 and 6 Day1
Plasma HDM201 concentration-time profiles | Cycle 1 Day 1, 2, 3, 8; Cycle 2, 3, 4, 5 and 6 Day 1
Plasma PK parameters of HDM201: AUC | Cycle 1 Day 1, 2, 3, 8; Cycle 2, 3, 4, 5 and 6 Day 1
Plasma PK parameters of HDM201: Cmax | Cycle 1 Day 1, 2, 3, 8; Cycle 2, 3, 4, 5 and 6 Day 1
Plasma PK parameters of HDM201: Tmax | Cycle 1 Day 1, 2, 3, 8; Cycle 2, 3, 4, 5 and 6 Day 1
Plasma PK parameters of HDM201: t1/2 | Cycle 1 Day 1, 2, 3, 8; Cycle 2, 3, 4, 5 and 6 Day 1
Plasma LXS196 concentration-time profiles in combination with HDM201 | Cycle 1 Day 1, 2, 3, 8; Cycle 2, 3, 4, 5 and 6 Day1
Plasma PK parameters of LXS196 in combination with HDM201:AUC | Cycle 1 Day 1, 2, 3, 8; Cycle 2, 3, 4, 5 and 6 Day1
Plasma PK parameters of LXS196 in combination with HDM201: Cmax | Cycle 1 Day 1, 2, 3, 8; Cycle 2, 3, 4, 5 and 6 Day1
Plasma PK parameters of LXS196 in combination with HDM201: Tmax | Cycle 1 Day 1, 2, 3, 8; Cycle 2, 3, 4, 5 and 6 Day1
Plasma PK parameters of LXS196 in combination with HDM201: t1/2 | Cycle 1 Day 1, 2, 3, 8; Cycle 2, 3, 4, 5 and 6 Day1
Plasma PK parameters of LXS196 in combination with HDM201: Racc | Cycle 1 Day 1, 2, 3, 8; Cycle 2, 3, 4, 5 and 6 Day1
LXS196 plasma protein binding as a single agent | Cycle 1 Day 1, 2, 15, 16
LXS196 plasma protein content as a single agent | Cycle 1, 2, 3 and 4 Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Columbia University Medical Center, New York, New York, United States
- Novartis Investigative Site, Westmead, New South Wales, Australia
- Novartis Investigative Site, Paris, France
- Novartis Investigative Site, Leiden, Netherlands
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17977